CLINICAL TRIAL: NCT06381505
Title: In Vivo Evaluation of a CT-Compatible Retractor for Image Guided Trans-Oral Surgery
Brief Title: RetracTOR/ Retractor for Image Guided Trans-Oral Surgery
Status: Not yet recruiting | Type: Observational
Sponsor: Ryan J. Halter (Other)
Collaborators: Dartmouth College (Other)
Responsible Party: Sponsor-Investigator, Ryan J. Halter, Investigator and Regulatory Sponsor, Dartmouth-Hitchcock Medical Center
Organization: Dartmouth-Hitchcock Medical Center (Other)
Other Study IDs: STUDY02002103
Record Dates: First submitted 2024-04-17; First posted 2024-04-24 (Actual); Last update posted 2024-04-26 (Actual); Status verified 2024-04

CONDITIONS: Oral Cavity Disease
Keywords: retractor
MeSH Terms: conditions — Mouth Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- custom device- radiolucent retractor: Custom device-radiolucent retractor used during staging endoscopy.

SUMMARY:
This study aims to demonstrate that a polymer retractor functions the same as a standard metal retractor used during endoscopy and throat surgery. The retractor is the device that holds the mouth open so the surgeon can easily access the mouth and throat. For example, this study aims to confirm that the mouth is held open the same amount with a polymer retractor as it is with a metal retractor. Benchtop experiments have demonstrated that the metal and polymer retractor's function the same, and thus this study will use this in patients.

DETAILED DESCRIPTION:
This study will include four stages of data collection: 1) Subject history, 2) intraoperative surgical working volume (SWV) assessment with stereoendoscopy and standard-of-care metal retractor, 3) intraoperative surgical working volume assessment with stereoendoscopy and 3D-printed polymer retractor, 4) intraoperative surgical working volume assessment with CT-imaging and 3D-printed polymer retractor.

The investigators will conduct a comparative study examining differences in surgical exposure within the same patient when retraction is enabled through use of standard-of-care metal retractor vs. our 3D printed retractor. Patients to be recruited for the study will include those who present to the Head and Neck Tumor Clinic at Dartmouth-Hitchcock Medical Center (DHMC) with suspicious lesions identified in the oropharynx, hypopharynx or larynx. Currently the clinic sees about 20 patients per month that are scheduled for staging endoscopy in the operating room. Consent will be obtained from all participating subjects prior to participation.

All surgeries will be performed at the Center for Surgical Innovation. Prior to surgery a standard-of-care Feyh-Kastenbauer (FK) or Crowe-Davis (CD) metal retractor will be positioned in the mouth of the patient and stabilized in suspension. A standard-of-care stereo vision endoscope will capture images of the oral cavity so that a 3D volume of the surgical working volume (SWV) can be measured. The time to place the retractor and surgical working volume metrics based on stereovision derived oral-cavity volumes and inter-incisive distance (IID) will be recorded. The FK and/or CD retractor will then be removed and replaced with our custom 3d-printed radiolucent retractor. The time to place this retractor and surgical working volume metrics based on stereovision derived oral-cavity volumes and inter-incisive distance will be recorded. A single CT scan with IV contrast will be obtained with the retractor in place and suspended. The standard surgical procedure will commence following routine methods. Following surgery, a second set of surgical working volume metrics based on stereovision derived oral-cavity volumes and inter-incisive distance will be recorded.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis or suspected cancer the oral cavity, oropharynx, hypopharynx, or larynx requiring resection.
2. Undergoing staging endoscopy at DHMC
3. Ability to understand and the willingness to sign a written informed consent document.
4. Age ≥ 18 years old
5. For females of child bearing potential, a negative pregnancy evaluation per standard of care.

Exclusion Criteria:

1. Prisoners
2. Adults with impaired decision-making capacity
3. Any condition for which, in the opinion of the investigator, contraindicates study participation.
4. Procedures that use high temperature generating devices such as laser

   -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Clinical diagnosis or suspected cancer the oral cavity, oropharynx, hypopharynx, or larynx requiring resection.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2024-05-15 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Comparing intraoperative surgical working volume (SWV) of a radiolucent retractor (custom device) as compared to SWV of standard-of-care metal retractors. | 2024-2025
  Assessment of intraoperative surgical working volume (SWV) during stereoendoscopy using standard-of-care metal retractor as compared to the same assessment parameters using 3D-printed polymer retractor during stereoendoscopy. Assessments will also include intraoperative SWV with CT-imaging taken with 3D-printed polymer retractor.

CONTACTS AND LOCATIONS:
Overall Officials: Ryan J Halter, PhD, Principal Investigator — Dartmouth-Hitchcock, Lebanon
Locations (1):
- Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire, United States

IPD SHARING:
Plan to Share IPD: No